CLINICAL TRIAL: NCT04830774
Title: Natural History and Recurrence Rate of Atrial Fibrillation After the First, COVID-19-Related Atrial Arrhythmic Episode: A Prospective Evaluation Using Continuous Cardiac Rhythm Monitoring
Brief Title: Natural History of COVID-19-Related Atrial Fibrillation
Acronym: unCOVer-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TCAI-unCOVer1
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Atrial Fibrillation New Onset
Keywords: atrial fibrillation; COVID-19; natural history; stroke; loop recorder; cardiac implantable electronic device; remote monitoring
MeSH Terms: conditions — COVID-19; Atrial Fibrillation; Stroke | interventions — Defibrillators, Implantable

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 patients with new-onset AF (Other): Consecutive patients with a confirmed diagnosis of COVID-19 with a first clinical episode of AF at admission or during hospitalization.
  Interventions: Device: ILR, PMK, ICD

INTERVENTIONS:
Device: ILR, PMK, ICD — * Patients receive a newly implanted ILR, PMK, or ICD during COVID-19 hospitalization or within 30 days after hospital discharge and are followed by daily automated remote transmissions.
  * Patients have a previously implanted ILR, PMK, or ICD and are followed by daily automated remote transmissions

SUMMARY:
The unCOVer-AF prospective, multicenter registry aims at determining the natural history of atrial fibrillation (AF) via continuous cardiac rhythm monitoring in patients with a first arrhythmic episode during COVID-19 hospitalization.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is a novel coronavirus strain disease, which has rapidly spread worldwide with more than 100 million confirmed cases to date. COVID-19 is mainly characterized by respiratory symptoms; however, patients can exhibit a wide range of clinical manifestations, including cardiovascular complications. Among them, supraventricular and ventricular arrhythmias have been described in patients at different stages of disease severity. According to a recent study on 9564 COVID-19 patients, 17.6% developed AF during hospitalization, 65.7% of whom without a past arrhythmic history.

Several factors (e.g., hypoxia, systemic inflammatory response, myocardial injury) may interact with a preexisting substrate and act as a trigger for AF initiation. Nonetheless, the pathophysiology of COVID-19-related new-onset AF remains elusive. It is unknown whether the disease merely acts as a transient arrhythmia initiator or promotes long-term atrial electrophysiological and structural changes which may facilitate AF recurrence and progression.

Therefore, the investigators designed a multicenter, prospective registry to assess the natural history of AF via continuous cardiac rhythm monitoring (ILR, PMK, ICD) in patients with a first AF episode during COVID-19 hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years;
* Confirmed infection with SARS-CoV-2;
* Patients with a first clinical episode of AF ≥30 s at admission or during hospitalization for COVID-19;
* Patients with:

  1. implantation of an ILR, a PMK, or an ICD during COVID-19 hospitalization or within 30 days after hospital discharge, or
  2. an ILR, a PMK, or an ICD implanted before COVID-19 hospitalization.

Exclusion Criteria:

* History of AF or flutter irrespective of type;
* Moderate/severe mitral stenosis;
* Mechanical prosthetic heart valve(s);
* Kidney failure treated with permanent dialysis;
* Any condition (e.g. psychiatric illness, dementia) or situation, that in the investigators opinion could put the subject at significant risk, confound the study results, or interfere significantly with the subject participation in the study;
* Unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
AF Burden | 3 years
  AF burden is defined as cumulative duration of all AF episodes lasting ≥30 s from the first adjudicated AF episode onward, divided by total duration of monitoring.
AF Progression | 3 years
Time to adjudicated ischemic stroke/transient ischemic attack (TIA)/systemic arterial embolism | 3 years

SECONDARY OUTCOMES:
Composite of all-cause mortality, stroke and bleeding | 3 years
Time to adjudicated cardiovascular death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Domenico G Della Rocca, MD, Study Director — Texas Cardiac Arrhythmia Research Foundation; Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (12):
- United States (2):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas City, Kansas
  - Texas Cardiac Arrhythmia Institute, Austin, Texas
- Vrije Universiteit Brussel, Brussels, Belgium
- Italy (9):
  - Department of Cardiovascular/Respiratory Diseases, Nephrology, Anesthesiology, and Geriatric Sciences, Policlinico Umberto I, Sapienza University of Rome, Rome, Lazio
  - Cardiology Unit, ASST-Fatebenefratelli Sacco, Luigi Sacco University Hospital, Milan, Italy, Milan, Lombardy
  - Ospedale San Donato, Arezzo
  - Maria Cecilia Hospital, Cotignola
  - Universita' Vanvitelli, Napoli
  - ARNAS Ospedale Civico, Palermo
  - Università di Pisa, Pisa
  - Policlinico Gemelli, Roma
  - Ospedale San Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mountantonakis SE, Saleh M, Fishbein J, Gandomi A, Lesser M, Chelico J, Gabriels J, Qiu M, Epstein LM; Northwell COVID-19 Research Consortium. Atrial fibrillation is an independent predictor for in-hospital mortality in patients admitted with SARS-CoV-2 infection. Heart Rhythm. 2021 Apr;18(4):501-507. doi: 10.1016/j.hrthm.2021.01.018. Epub 2021 Jan 22. PMID 33493650